CLINICAL TRIAL: NCT04074057
Title: Effectiveness of a Novel Mobile App Based Cardiac Rehabilitation Compared to Traditional Centre-based, Therapist Driven Cardiac Rehabilitation for Patients Post Coronary Revascularisation : A Non-inferiority Pilot Study
Brief Title: Effectiveness of a Novel Mobile App Based Cardiac Rehabilitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tan Tock Seng Hospital (Other)
Responsible Party: Principal Investigator, Eng Chan Neoh, Senior Physiotherapist, Tan Tock Seng Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018/00977
Record Dates: First submitted 2019-08-20; First posted 2019-08-29 (Actual); Last update posted 2019-08-29 (Actual); Status verified 2019-08

CONDITIONS: Cardiac Disease
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Intervention Model Description: All patients who are referred for Cardiac Rehabilitation post discharge from hospital will be assessed by the Physiotherapist during the first follow-up appointment to determine eligibility for inclusion. During this session, exercise testing and a body composition analysis will be done for every patient. The Physiotherapist will then stratify all patients into low, moderate and high-risk groups only those with low and moderate risk will be included into the study after informed consent is attained. A research assistant randomise the patients into two groups, namely the intervention group or the control group. Block randomisation method will be used by using the randomisation function in Red Cap created by independent aata manager who is not part of the study team.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Randomization and group allocation are done by the research coordinator. Final assessment is also arranged by research coordinator. Blinded assessor will conduct the final assessment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (Other): the control group will undergo a conventional weekly CR programme lasting 8-12 sessions. Components of each session will include warm up, aerobic training, resistance exercises and cool down. Patients are encouraged to continue their home exercises, exercising another 2 times a week at home and record down using an activity diary. The importance of CR programme and exercise advice will be explained and reinforced by the CR Physiotherapist. The submaximal exercise test and a body composition analysis will be repeated on the final assessment. Every week research coordinator will call the subject to remind them to exercise.
  Interventions: Other: Conventional Cardiac Rehab Classes
- Intervention arm (Other): During the initial assessment, the importance of CR and regular exercise will be explained and reinforced by CR physiotherapist. A research assistant will teach the patient how to use "Heart Track". The patient will then bring "Heart Track" home to continue their CR program. Patient will then undergo the whole CR programme to exercise for 3 times a day for 8-12 weeks using "Heart Track". Each "Heart Track" session will include warm up, aerobic training, resistance exercises and cool down (same as the traditional CR session). After 8-12 weeks, patient will be called back to the clinic by the research assistant to complete the final assessment (sub-maximal exercise test and a body composition analysis) with the blinded assessor. Every week research coordinator will call the subject to remind them to exercise.
  Interventions: Device: Heart Track

INTERVENTIONS:
Other: Conventional Cardiac Rehab Classes — conventional weekly CR programme lasting 8-12 sessions.
  Arms: Control arm
Device: Heart Track — Key components of "Heart-Track" are a heart rate sensor, a mobile app and a remote monitoring portal. The "Heart-Track" mobile app is synchronized/ connected to Polar heart rate sensor through bluetooth in order to provide continous heart rate monitoring when subjects are exercising. This is to ensure safety and exercise effectiveness.
  Arms: Intervention arm

SUMMARY:
n Tan Tock Seng (TTSH), Acute myocardial infarction (AMI) is one of the top 4 reasons for admissions with 948 percutaneous coronary intervention (PCI) procedures done in year 2016. International guidelines recommend that all patients complete CR after PCI, as it plays a critical role in reducing five-year cardiovascular mortality and the risk of cardiovascular-related hospital admission. However, the rate of completion of CR has been found to be low as only 19% of post PCI patients completed CR in 2016. According to a patient survey conducted, the main reason for non-completion is the inconvenience experienced by patients from needing to return to hospital weekly. In addition, poor compliance to prescribed home exercises limits the effectiveness of exercise training. Hence, there is a pertinent need to activate patients to engage in self-directed CR in a safe and effective manner to target these issues. Current solutions to increase participation and compliance involve strategies have been limited. Participation and compliance to prescribed exercises recorded via brochures and activity diaries have been limited by difficulties experienced by patients when providing this information, posing a risk of recall bias or the risk of misplacing their activity logs. Mobile applications targeted at increasing fitness addresses the problem of the risk of misplacing activity logs but is still subjected to recall bias as self-input of multiple data is required. Exercise guidelines within these applications are also generic and does not adhere to international exercise training guidelines targeted at patients after coronary revascularisation. In order to address these gaps, there is a need for a technology enabled solution that can provide evidence-based CR programme with constant HR monitoring which offers direct feedback to the patients and at the same time affordable and easy to use. "Heart-Track" is a novel mobile app based CR model of care that utilises a technology-enabled device designed specifically for patients post PCI to complete CR at their convenience, while ensuring that evidence-based clinical outcomes are achieved.

DETAILED DESCRIPTION:
In Tan Tock Seng (TTSH), Acute myocardial infarction (AMI) is one of the top 4 reasons for admissions with 948 percutaneous coronary intervention (PCI) procedures done in year 2016. International guidelines recommend that all patients complete CR after PCI, as it plays a critical role in reducing five-year cardiovascular mortality and the risk of cardiovascular-related hospital admission. However, the rate of completion of CR has been found to be low as only 19% of post PCI patients completed CR in 2016. According to a patient survey conducted, the main reason for non-completion is the inconvenience experienced by patients from needing to return to hospital weekly. In addition, poor compliance to prescribed home exercises limits the effectiveness of exercise training. Hence, there is a pertinent need to activate patients to engage in self-directed CR in a safe and effective manner to target these issues. Current solutions to increase participation and compliance involve strategies have been limited. Participation and compliance to prescribed exercises recorded via brochures and activity diaries have been limited by difficulties experienced by patients when providing this information, posing a risk of recall bias or the risk of misplacing their activity logs. Mobile applications targeted at increasing fitness addresses the problem of the risk of misplacing activity logs but is still subjected to recall bias as self-input of multiple data is required. Exercise guidelines within these applications are also generic and does not adhere to international exercise training guidelines targeted at patients after coronary revascularisation. In order to address these gaps, there is a need for a technology enabled solution that can provide evidence-based CR programme with constant HR monitoring which offers direct feedback to the patients and at the same time affordable and easy to use. "Heart-Track" is a novel mobile app based CR model of care that utilises a technology-enabled device designed specifically for patients post PCI to complete CR at their convenience, while ensuring that evidence-based clinical outcomes are achieved. The key components of "Heart-Track" are: 1. Exercise principles based on international guidelines 2. Gamification; 3. Continuous heart rate monitoring; 4. Adaptation to local context. As Heart-track is the first of its kind, being designed for use in the local context, findings from research is important in determining its efficacy when compared to traditional cardiac rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

1. 21-65 years old
2. Underwent coronary revascularisation follow AMI
3. Language literacy English or Mandarin
4. Owns a smart phone
5. Normal physiological response during exercise testing
6. Low or moderate risk following risk stratification.

Exclusion Criteria:

1. Medically unfit for exercise
2. Post op complication
3. High risk following risk stratification
4. Cognitive impaired

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-05-31 (Estimated); Study Completion 2020-05-31 (Estimated)

PRIMARY OUTCOMES:
6 minutes walk test | through study completion, an average of 1 year
  The 6-min walk test (6 MWT) is a submaximal exercise test that entails measurement of distance walked over a span of 6 minutes. The MCID for 6MWD in patients with CAD after ACS was 25m.
Body weight | through study completion, an average of 1 year
  Body weight will be assessed , record in kg
Body Height | through study completion, an average of 1 year
  Body height will be assessed, record in meter
Body Mass Index | through study completion, an average of 1 year
  Measure of body fat based on height and weight that applies to adult men and women. Calculated by using body weight and height (kg/m2)
Body Fat Percentage | through study completion, an average of 1 year
  Assess using a bioelectrical impedance analysis (BIA) method, record in percentage %
Skeletal muscle mass | through study completion, an average of 1 year
  Assess using a bioelectrical impedance analysis (BIA) method, record in kg
Waist Hip Ratio | through study completion, an average of 1 year
  Assess using a bioelectrical impedance analysis (BIA) method
Borg's RPE scale | through study completion, an average of 1 year
  Rating of perceived exertion (RPE) is a widely used and reliable indicator to monitor and guide exercise intensity. The scale allows individuals to subjectively rate their level of exertion during exercise or exercise testing. body fat,Skeletal muscle mass, Waist-hip ratio can be measured by using the body composition analysis machine. Borg scale 6-20, 6 is very very light and 20 is very very hard.

SECONDARY OUTCOMES:
Self-Efficacy for Exercise Scale• | through study completion, an average of 1 year
  This scale is a self-report of exercise self-efficacy. Total score is calculated by summing the responses to each question. This scale has a range of total scores from 0-90. A higher score indicates higher self-efficacy for exercise.
Health related QoL: MacNew myocardial infarction Quality of life questionnaire | through study completion, an average of 1 year
  1. The MacNew consists of 27 items which fall into three domains [a 13-item physical limitations domain scale, a 14-item emotional function domain scale, and a 13-item social function domain scale]. There are 5 items that inquire about symptoms: angina/chest pain, shortness of breath, fatigue, dizziness, and aching legs.
  2. Scores are reported using a descriptive scale which are described as: "all of the time", "most of the time", "a good bit of the time", "some of the time", "a little of the time", "hardly any of the time" and "none of the time"
  3. The maximum possible score in any domain is 7 [high HRQL] and the minimum is 1 [poor HRQL]
Patient-reported survey on usability of Heart Track acceptability | through study completion, an average of 1 year
  Participants rated their experience with the hardware and software components of "Heart Track", and their acceptance of it as a cardiac rehabilitation tool. The survey form is a likert-scale ( Strongly agree to strongly disagree) survey that asking subjects about their feedback and satisfaction about the Heart Track hardware and software, and overall experience using Heart Track.

CONTACTS AND LOCATIONS:
Overall Officials: Eng Chuan Neoh, masters, Study Director — Senior Physiotherapist
Locations (1):
- Tan Tock Seng Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No